CLINICAL TRIAL: NCT01851538
Title: Serial Biomarker Measurements and New Echocardiographic Techniques in Chronic Heart Failure Patients Result in Tailored Prediction of Prognosis
Brief Title: The Role of Biomarkers and Echocardiography in Prediction of Prognosis of Chronic Heart Failure Patients
Acronym: Bio-SHiFT
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, Eric Boersma, Prof.dr., Erasmus Medical Center
Other Study IDs: MEC-2011-029
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Biomarkers; Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (EDTA plasma, citrate plasma, serum, DNA) and urine samples are taken at the day of inclusion and at follow-up visits, which will be performed every 3 months, until the end of the scheduled follow-up, or until the patient dies. The maximum total number of samples per patient is 11 (in patients with 30 months follow-up).

GROUPS / COHORTS (1):
- Chronic heart failure patients visiting the outpatient clinic
  Interventions: Other: Observational study; no intervention.

INTERVENTIONS:
Other: Observational study; no intervention.

SUMMARY:
The Bio-SHiFT study aims to investigate whether disease progression in individual patients with chronic heart failure (CHF) can be accurately assessed by serial measurements of disease-related (novel) biomarkers. Secondary objectives of the study include comparison of 2D- with real-time 3D-echocardiography in CHF patients and comparison of Speckle tracking with tissue Doppler imaging (TDI) in CHF patients, and relating these echocardiographic measurements to clinical outcome.

Bio-SHiFT is a prospective, observational, multi-center, cohort study in men and women, aged 18 years or older, visiting the outpatient clinic. Blood samples are taken at the day of inclusion and at follow-up visits, which are performed every 3 months until the end of the scheduled follow-up. Clinical data are collected at baseline and at each 3-month follow-up visit. Echocardiography including TDI, Speckle tracking and 3D-echocardiography is performed in a subset of patients, at baseline and during follow-up at 6-month intervals. The primary endpoint is the composite of cardiovascular death, cardiac transplantation, left ventricular assist device implantation, and re-hospitalization for the management of acute or worsened heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years or older, capable of understanding and signing informed consent
* Diagnosis of chronic heart failure (with diminished ejection fraction or with normal ejection fraction), according to the guidelines of the European Society of Cardiology (ESC)

Exclusion Criteria:

* Heart failure secondary to circulatory high output conditions
* Scheduled for surgery or intervention for both coronary and non-coronary indication
* Severe renal failure for which dialysis is needed
* Known moderate or severe liver disease
* Chronic Obstructive Pulmonary Disease (COPD) Gold stage IV
* Congenital heart disease
* Coexistent condition with life expectancy ≤ 1 year
* Unlikely to appear at all scheduled follow-up visits
* Linguistic barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic heart failure patients visiting the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2011-08; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
The composite of cardiovascular death, cardiac transplantation, left ventricular assist device implantation, and re-hospitalization for the management of acute or worsened heart failure. | maximum follow-up is 2.5 years

SECONDARY OUTCOMES:
Cardiovascular death | maximum follow-up is 2.5 years
Cardiac transplantation | maximum follow-up is 2.5 years
Left ventricular assist device implantation | maximum follow-up is 2.5 years
Re-hospitalization for acute or worsened heart failure | maximum follow-up is 2.5 years
Cardiovascular disease: myocardial infarction (fatal and non-fatal), stroke (fatal and non-fatal), percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG) | maximum follow-up is 2.5 years
  Cardiovascular disease, comprising all events specified above, will be examined, as well as all individual components.
All-cause mortality | maximum follow-up is 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boersma, MSc, PhD, Study Chair — Erasmus Medical Center; Isabella Kardys, MD, PhD, Study Director — Erasmus Medical Center; Victor Umans, MD, PhD, Principal Investigator — Medical Center Alkmaar; Martijn Akkerhuis, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Medical Center Alkmaar, Alkmaar
  - Erasmus MC, Rotterdam

REFERENCES:
- [Derived] de Bakker M, Petersen TB, Rueten-Budde AJ, Akkerhuis KM, Umans VA, Brugts JJ, Germans T, Reinders MJT, Katsikis PD, van der Spek PJ, Ostroff R, She R, Lanfear D, Asselbergs FW, Boersma E, Rizopoulos D, Kardys I. Machine learning-based biomarker profile derived from 4210 serially measured proteins predicts clinical outcome of patients with heart failure. Eur Heart J Digit Health. 2023 Oct 4;4(6):444-454. doi: 10.1093/ehjdh/ztad056. eCollection 2023 Dec. PMID 38045440
- [Derived] Petersen TB, de Bakker M, Asselbergs FW, Harakalova M, Akkerhuis KM, Brugts JJ, van Ramshorst J, Lumbers RT, Ostroff RM, Katsikis PD, van der Spek PJ, Umans VA, Boersma E, Rizopoulos D, Kardys I. HFrEF subphenotypes based on 4210 repeatedly measured circulating proteins are driven by different biological mechanisms. EBioMedicine. 2023 Jul;93:104655. doi: 10.1016/j.ebiom.2023.104655. Epub 2023 Jun 14. PMID 37327673
- [Derived] Klimczak-Tomaniak D, de Bakker M, Bouwens E, Akkerhuis KM, Baart S, Rizopoulos D, Mouthaan H, van Ramshorst J, Germans T, Constantinescu A, Manintveld O, Umans V, Boersma E, Kardys I. Dynamic personalized risk prediction in chronic heart failure patients: a longitudinal, clinical investigation of 92 biomarkers (Bio-SHiFT study). Sci Rep. 2022 Feb 18;12(1):2795. doi: 10.1038/s41598-022-06698-3. PMID 35181700
- [Derived] Bouwens E, Schuurman AS, Akkerhuis KM, Manintveld OC, Caliskan K, van Ramshorst J, Germans T, Umans VA, Boersma E, Kardys I. Associations of serially measured PCSK9, LDLR and MPO with clinical outcomes in heart failure. Biomark Med. 2021 Mar;15(4):247-255. doi: 10.2217/bmm-2020-0585. Epub 2021 Feb 16. PMID 33590771
- [Derived] Bouwens E, Brankovic M, Mouthaan H, Baart S, Rizopoulos D, van Boven N, Caliskan K, Manintveld O, Germans T, van Ramshorst J, Umans V, Akkerhuis KM, Kardys I. Temporal Patterns of 14 Blood Biomarker candidates of Cardiac Remodeling in Relation to Prognosis of Patients With Chronic Heart Failure-The Bio- SH i FT Study. J Am Heart Assoc. 2019 Feb 19;8(4):e009555. doi: 10.1161/JAHA.118.009555. PMID 30760105